CLINICAL TRIAL: NCT03285308
Title: A 12-week, Randomized, Double-blind, Placebo-controlled, Phase 3 Study to Evaluate the Safety and Efficacy of Relamorelin in Patients With Diabetic Gastroparesis
Brief Title: A Safety and Efficacy Study of Relamorelin in Diabetic Gastroparesis 01
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The Relamorelin program is being terminated solely based on a business decision.
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RLM-MD-01; 2017-002136-16 (EudraCT Number)
Record Dates: First submitted 2017-09-14; First posted 2017-09-18 (Actual); Results first posted 2021-07-29 (Actual); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Gastroparesis; Diabetes Mellitus
MeSH Terms: conditions — Gastroparesis; Diabetes Mellitus | interventions — relamorelin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Following a 2-week placebo run-in, participants received placebo-matching relamorelin injected subcutaneously twice daily for up to 12 weeks.
  Interventions: Drug: Placebo
- Relamorelin 10 μg (Experimental): Following a 2-week placebo run-in, participants received relamorelin 10 μg injected subcutaneously twice daily for up to 12 weeks.
  Interventions: Drug: Relamorelin

INTERVENTIONS:
Drug: Placebo — Placebo injected subcutaneously twice daily.
  Arms: Placebo
Drug: Relamorelin — Relamorelin 10 micrograms (μg) injected subcutaneously twice daily.
  Arms: Relamorelin 10 μg

SUMMARY:
This study will evaluate the safety and efficacy of relamorelin compared to placebo in participants with diabetic gastroparesis. Participants will report daily severity scores of their diabetic gastroparesis symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Type 1 or Type 2 diabetes mellitus
* Meet the per protocol criteria of diabetic gastroparesis
* Compliance with diary
* Compliance with the per protocol study treatment dosing instructions

Exclusion Criteria:

* Currently receiving nutrition intravenously, by nasogastric tube, or other feeding tube
* Actively experiencing anorexia nervosa, binge-eating, bulimia, or other eating disorder at the time of Screening (Visit 1)
* Diagnosis of Celiac Disease, also a history of non-celiac gluten sensitivity
* History of gastrointestinal disorders that may be similar to gastroparesis
* Functional dyspepsia diagnosed before the diagnosis of diabetes mellitus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 336 (Actual)
Dates: Start 2017-09-29 (Actual); Primary Completion 2020-07-08 (Actual); Study Completion 2020-07-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wieslaw (Wes) Bochenek, MD, PhD, Study Director — Allergan
Locations (216):
- United States (113):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Digestive Health Specialist of the South East, Dothan, Alabama
  - Avant Research Associates, Huntsville, Alabama
  - Synexus Clinical Research US, Inc., Fountain Hills, Arizona
  - Central Arizona Medical Associates, Mesa, Arizona
  - Phoenix Clinical LLC, Phoenix, Arizona
  - Del Sol Research Management, LLC, Tucson, Arizona
  - Preferred Research Partners, Inc., Little Rock, Arkansas
  - Arkansas Gastorenterology, North Little Rock, Arkansas
  - Hope Clinical Research, Canoga Park, California
  - Kindred Medical Institute for Clinical Trials, LLC, Corona, California
  - Aurora Care Clinic, LLC, Costa Mesa, California
  - Citrus Valley Gastroenterology Clinic, Covina, California
  - VVCRD Research, Garden Grove, California
  - University of California San Diego, La Jolla, California
  - Om Research LLC, Lancaster, California
  - Clinical Applications Laboratories, Inc., San Diego, California
  - Medical Associates Research Group, Inc, San Diego, California
  - Synexus Clinical Research, US, Santa Rosa, Santa Rosa, California
  - Upland Clinical Research, Upland, California
  - Synexus Clinical Research US, Inc., Vista, California
  - University of Colorado, Denver, Aurora, Colorado
  - Peak Gastroenterology Associates, Colorado Springs, Colorado
  - Denver Esophageal and Stomach Center, Englewood, Colorado
  - Connecticut Clinical Research Foundation, Bristol, Connecticut
  - Medical Research Center of Connecticut, LLC, Hamden, Connecticut
  - TrialSpark, Inc., Washington D.C., District of Columbia
  - Innovative Research of West FL, Inc., Clearwater, Florida
  - West Central Gastroenterology, Clearwater, Florida
  - American Research Institute, Inc, Cutler Bay, Florida
  - Top Medical Research, Cutler Bay, Florida
  - Nature Coast Clinical Research, Inverness, Florida
  - Cfagi Llc, Maitland, Florida
  - APF Research LLC, Miami, Florida
  - AMPM Research Clinic, Miami, Florida
  - Advanced Medical Research Institute, Miami, Florida
  - Florida Research Center, Inc., Miami, Florida
  - Savin Medical Group LLC, Miami Lakes, Florida
  - Sensible Healthcare, Ocoee, Florida
  - Gulf Region Clinical Research Institute, Pensacola, Florida
  - University of South Florida, Tampa, Florida
  - West Central Gastroenterology, Tampa, Florida
  - Summit Clinical Research, LLC, Carnesville, Georgia
  - Infinite Clinical Trials, Riverdale, Georgia
  - Southwest Gastroenterology, Oak Lawn, Illinois
  - MediSphere Medical Research Center, LLC, Evansville, Indiana
  - Synexus Clinical Research US, Inc., Evansville, Indiana
  - Indiana University Health University Hospital, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Cotton-O'Neil Clinical Research Center - Digestive Health, Topeka, Kansas
  - University of Louisville, Louisville, Kentucky
  - Delta Research Partners, Bastrop, Louisiana
  - Cronola LLC, Houma, Louisiana
  - New Orleans Research Institute - Metropolitan Gastroenterology Associates, Metairie, Louisiana
  - Gastro Center of Maryland, Columbia, Maryland
  - Frederick Gastroenterology Associates, PA an Elligo Health Research Site, Frederick, Maryland
  - Boston VA Healthcare System, West Roxbury, Massachusetts
  - Vida Clinical Studies, Dearborn, Michigan
  - National Clinical, LLC, Hamtramck, Michigan
  - Henry Ford Health System, Novi, Michigan
  - Gastroenterology Associates of Western Michigan, Wyoming, Michigan
  - MNGI Digestive Health, Coon Rapids, Minnesota
  - Synexus Clinical Research US, Inc., Richfield, Minnesota
  - Montana Medical Research, Missoula, Montana
  - Synexus Clinical Research, Henderson, Nevada
  - Excel Clinical Research, Las Vegas, Nevada
  - Clinical Research of South Nevada, Las Vegas, Nevada
  - Advanced Biomedical Research of America, Las Vegas, Nevada
  - Digestive Disease Specialists, Las Vegas, Nevada
  - Palm Research Center, Las Vegas, Nevada
  - Garden State Endocrinology, Brick, New Jersey
  - Synexus Clinical Research US, Inc., Bridgeton, New Jersey
  - AGA Clinical Research Associates LLC, Egg Harbor, New Jersey
  - Long Island Gastrointestinal Research Group LLP, Great Neck, New York
  - United Health Services Hospitals, Inc., Johnson City, New York
  - CHEAR Center, LLC, The Bronx, New York
  - Asheville Gastroenterology Associates, Asheville, North Carolina
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Carolinas Healthcare-Charlotte, Charlotte, North Carolina
  - Carolina Digestive Health Associates, Concord, North Carolina
  - Cumberland Research Associates, LLC, Fayetteville, North Carolina
  - Triad Clinical Trials, Greensboro, North Carolina
  - PMG Research Salisbury, Salisbury, North Carolina
  - The Center for Clinical Research, Winston-Salem, North Carolina
  - Dayton Gastroenterology,Inc., Beavercreek, Ohio
  - Endocrinology Research Associates, Inc., Columbus, Ohio
  - Hometown Urgent Care and Research, Columbus, Ohio
  - Premier Clinical Research d.b.a. STAT Research, Franklin, Ohio
  - Family Practice Center of Wadsworth, Inc., Wadsworth, Ohio
  - Digestive Disease Specialists Inc, Oklahoma City, Oklahoma
  - Memorial Clinical Research, Oklahoma City, Oklahoma
  - Northwest Gastroenterology Clinic, LLC, Portland, Oregon
  - Family Medical Associates, Research Department, Levittown, Pennsylvania
  - Preferred Primary Care Physicians, Inc., Pittsburgh, Pennsylvania
  - Montgomery Medical, Inc., Smithfield, Pennsylvania
  - Synexus Clinical Research US, Inc., Anderson, South Carolina
  - Carolina Medical Research, Clinton, South Carolina
  - Gastroenterology Associates, PA, Greenville, South Carolina
  - Synexus Clinical Research, Greer, South Carolina
  - Quality Medical Research, Nashville, Tennessee
  - Avant Research Associates,LLC, Austin, Texas
  - Synexus Clinical Research US, Inc., Dallas, Texas
  - Amir Ali Hassan, MD, PA, Houston, Texas
  - Clinical Trials of Texas, Inc., San Antonio, Texas
  - Sagact Pllc, San Antonio, Texas
  - Synexus Clinical Research US, Inc., Layton, Utah
  - Synexus Clinical Research US, Inc., Murray, Utah
  - Advanced Research Institute, Inc., Ogden, Utah
  - Advanced Clinical Research, West Jordan, Utah
  - Verity Research Inc., Fairfax, Virginia
  - Cardinal Internal Medicine, Woodbridge, Virginia
  - West Virginia University, Morgantown, West Virginia
- Australia (4):
  - Nepean Hospital, Kingswood, New South Wales
  - Royal Adelaide Hospital - Central Adelaide Local Health Network Incorporated, Adelaide, South Australia
  - The Alfred Hospital, Melbourne, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
- Bulgaria (4):
  - MHAT Yuliya Vrevska Byala, Byala, Ruse
  - UMHAT - Kaspela- EOOD, Plovdiv
  - Medical Center Asklepion - Humane Medicine Research EOOD, Sofia
  - Alexandrovska University Hospital, Sofia
- France (2):
  - CHU Nantes, Nantes
  - Hopital Charles Nicolle, Rouen
- India (22):
  - Kumudini Devi Diabetes Research Center; Ramdevrao Hospital, Hyderabad, Andhra Pradesh
  - King George Hospital, Visakhapatnam, Andhra Pradesh
  - Dr. Jivraj Mehta Smarak Health Foundation Bakeri Medical Research Centre - Gasterentrology, Ahmedabad, Gujarat
  - Victoria Hospital, Bangalore, Karnataka
  - Life Care Hospital & Research Centre, Bangalore, Karnataka
  - Diacon Hospital and research Center - Diabetology, Bengaluru, Karnataka
  - Rajalakshmi Hospital, Bengaluru, Karnataka
  - Vinaya Hospital & Research Centre, Mangalore, Karnataka
  - Bhatia Hospital, Mumbai, Maharashtra
  - B. J. Government Medical College and Sassoon General Hospitals, Pune, Maharashtra
  - Universal Hospital, Pune, Maharashtra
  - Noble Hospital Pvt. Ltd, Pune, Maharashtra
  - S R Kalla (SRK) Memorial Gastro & General Hospital, Jaipur, Rajasthan
  - SMS Hospital, Jaipur, Rajasthan
  - Diabetic Thyroid and Endocrine Centre, Jaipur, Rajasthan
  - Marudhar Hospital, Jaipur, Rajasthan
  - Eternal Hospital - Diabetology, Jaipur, Rajasthan
  - M.V. Hospital for Diabetes & Diabetes Research Centre, Chennai, Tamil Nadu
  - Kovai Diabetes Speciality Centre, Coimbatore, Tamil Nadu
  - M V Hospital & Research Centre, Lucknow, Uttar Pradesh
  - Arthur Asirvatham Hospital, Madurai
  - Sir Ganga Ram Hospital, New Delhi
- Israel (7):
  - Soroka University Medical Center, Beersheba
  - Bnai Zion Medical Center, Haifa
  - E. Wolfson Medical Center, Holon
  - Digestive Diseases Institute, Jerusalem
  - Gastroenterology Institute, Petah Tikva
  - Endocrinology & Diabetes Center, Safed
  - Gastroenterology Institute, Tel Aviv
- Malaysia (4):
  - Hospital Sultanah Bahiyah, Alor Star, Kedah
  - University Malaya Medical Centre, Kuala Lumpur
  - Universiti Sains Malaysia, Kubang Kerian
  - Hospital Taiping, Taiping
- Philippines (7):
  - Manila Doctors Hospital, Ermita, Manila
  - San Juan De Dios Educational Foundation, Inc., Pasay, National Capital Region
  - Cardinal Santos Medical Center, San Juan City, National Capital Region
  - Ospital ng Makati, Makati City, NCR
  - Perpetual Succor Hospital, Cebu City
  - West Visayas State University Medical Center, Iloilo City
  - St. Luke's Medical Center, Quezon City
- Poland (15):
  - Synexus Polska Sp.z o.o., Pomorskie, Gdansk
  - CenterMed Krakow Ltd, Krakow, Malopolska
  - Centrum Medyczne Pratia S.A. Warsaw, Poland, Warsaw, Mazowian
  - Endoskopia Sp. Z O.O., Sopot, Pomeranian Voivodeship
  - Synexus Polska Sp. z o.o.Oddzial w Poznaniu, Poznan, Poznañ
  - Wojewodzki Szpital Specjalistyczny w Olsztynie, Olsztyn, Warmian-Masurian Voivodeship
  - NZOZ Vita Diabetica - Malgorzata Buraczyk, Bialystok
  - Centrum Medyczne Lukamed, Chojnice
  - Synexus Polska sp.z.o.o oddzial Czestochowa, Częstochowa
  - Specjalistyczny Gabinet Neurologiczny Marta Banach, Krakow
  - Synexus Polska Sp. z o.o. Oddzial w Lodzi, Lodz
  - Sanitas Centrum Medyczne, Lublin
  - Synexus Polska Sp. z o.o. Oddzial w Warszawie, Warsaw
  - DRS Wroclaw, Wroclaw
  - Centrum Badan Klinicznych Piotr Napora Lekarze Spolka Partnerska, Wroclaw
- Singapore (3):
  - National University Hospital, Singapore
  - Changi General Hospital, Singapore
  - Singapore General Hospital, Singapore
- South Korea (3):
  - Chonbuk National University Hospital, Jeonju, Jeollabuk-do
  - Sanggye Paik Hospital, Inje University College of Medicine, Seoul, Nowon-gu
  - Asan Medical Center, Seoul
- Spain (3):
  - Hospital Universitario Principe de Asturias, Madrid
  - Hospital Universitario De Salamanca, Salamanca
  - Hospital Universitario Virgen del Rocío, Seville
- Thailand (3):
  - Phramongkutklao Hospital, Bangkok
  - Faculty of Medicine, Siriraj Hospital, Mahidol University, Bangkok
  - Maharaj Nakorn Chiang Mai Hospital, Chiang Mai
- Ukraine (26):
  - Communal Institution "Odesa Regional Clinical Hospital", Out-patient department, Odesa, Odesa Oblast
  - Limited Liability Company "Medical Center "Salutem", Vinnitsa, Vinnytsia Oblast
  - Municipal Institution City Hospital No. 7, Zaporizhzhia, Zaporizhzhia Oblast
  - Regional municipal institution "Chernivtsi's regional clinical hospital", gastroenterological department, Higher state educational establishment of Ukraine "Bukovinian state medical university", department of internal medicine and infectious diseases, c.C, Chernivtsi
  - Regional Public Organization Chernivtsi Regional Endocrinology Center, Chernivtsi
  - State Institution Ukrainian State Research Institute of Medical and Social Problems of Disability of the Ministry of Health of Ukraine, Dnipro
  - Ivano-Frankivsk National Medical University, Ivano-Frankivsk
  - Ivano-Frankivsk Central City Clinical Hospital, Ivano-Frankivsk
  - Municipal nonprofit entity of Kharkiv municipal council, Kharkiv
  - L.T.Malaya Therapy National Institute of the National Academy of Medical Sciences of Ukraine, Kharkiv
  - Clinical Endocrinology of SI "V.Danilevsky Institute for endocrine pathology problems National Academy of Medical sciences of Ukraine", Kharkiv
  - Communal Institution Kherson City Clinical Hospital, Kherson
  - Kyiv municipal clinical endocrinological center, Kyiv
  - AS Medbud Clinic, Kyiv
  - AS PVNZ, Kyiv
  - Limited Liability Company "Medical and Diagnostic Center "ADONIS Plus", outpatient department, c. Kyiv, Kyiv
  - Kyiv Railway hospital on the railway transport #2 of the branch "health, Kyiv
  - Medical Center Universal Clinic Oberig, Kyiv
  - Polyclinic of medical services and rehabilitation department of State Joint-Stock Holding Company Artem, day-patient unit, Kyiv
  - Odessa Railway Clinical Hospital of Branch of HC JSC Ukrzaliznytsia, Odessa National Medical University, Odesa
  - Poltava Regional Clinical Hospital, Poltava
  - Ternopil University Hospital, Ternopil
  - Private Small-Scale Enterprise Medical Centre Pulse, Vinnytsia
  - Vinnytsia Regional Clinical highly specialized Endocrinology Centre, Vinnytsia
  - Municipal nonprofit entity "Vinnytsia's city clinical hospital #1", c. Vinnytsia, Vinnytsia
  - 6th City Clinical Hospital, c. Zaporizhzhia, Zaporizhzhia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Relamorelin 10 μg
Started | 167 | 169
Safety Population (Safety Population included participants who received ≥1 administration of Double-blind study treatment.) | 163 | 163
Completed | 147 | 146
Not Completed | 20 | 23
Not completed — Adverse Event | 3 | 7
Not completed — Withdrawal by Subject | 8 | 9
Not completed — Lost to Follow-up | 3 | 1
Not completed — Protocol Deviation | 6 | 5
Not completed — Reason not Specified | 0 | 1

BASELINE CHARACTERISTICS:
Population: ITT Population included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Relamorelin 10 μg | Total
Number analyzed (Participants) | 167 | 169 | 336
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.4 (10.78) | 56.3 (11.47) | 55.9 (11.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 107 | 115 | 222
  Male | 60 | 54 | 114
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 51 | 53 | 104
  Not Hispanic or Latino | 116 | 116 | 232
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 26 | 24 | 50
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 25 | 19 | 44
  White | 116 | 125 | 241
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 12 in the Weekly Diabetic Gastroparesis Symptom Severity Score (DGSSS)
Description: Participants assessed the severity of diabetic gastroparesis symptoms daily using the Diabetic Gastroparesis Symptom Severity Diary (DGSSD), recorded in an electronic diary (e-diary). The DGSSS was derived as the sum of the weekly averages of the 4 DGSSD items: nausea, abdominal pain, postprandial fullness and bloating. Each symptom was scored using an 11-point ordinal scale where: 0=no or not at all uncomfortable to 10=worst possible or most uncomfortable for a total possible DGSSS of 0 (best) to 40 (worst). A negative change from Baseline indicates improvement. Baseline was defined as the average of the 2 weekly DGSSS from the Run-in Period.
Time Frame: Baseline (Day-14 to Day-1) to Week 12
Population: Modified Intent-to-treat (mITT) Population included all randomized participants with ≥1 postbaseline assessment of DGSSD. Number analyzed is the number of participants with data available at the given time-point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Relamorelin 10 μg
Number analyzed (Participants) | 163 | 165
score on a scale
  Baseline | 25.1 (5.53) | 24.5 (5.99)
  Change from Baseline to Week 12: number analyzed (Participants) | 142 | 141
  Change from Baseline to Week 12 | -10.0 (8.89) | -9.3 (8.17)

2. Primary Outcome: Percentage of Participants Meeting the Vomiting Responder Criterion During Each of the Last 6 Weeks of the 12-week Treatment Period
Description: The number of vomiting episodes in the previous 24 hours were assessed daily by the participant using the DGSSD and were recorded in the e-diary. A Vomiting Responder was defined as a participant with zero weekly vomiting episodes during each of the last 6 weeks of the 12-week Treatment Period.
Time Frame: Week 6 to Week 12
Population: mITT Population included all randomized participants with ≥1 postbaseline assessment of DGSSD.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Relamorelin 10 μg
Number analyzed (Participants) | 164 | 165
percentage of participants | 19.5 | 21.8

3. Secondary Outcome: Percentage of Participants Meeting the Nausea Responder Criterion During Each of the Last 6 Weeks of the 12-week Treatment Period
Description: A Nausea Responder was defined as a participant with improvement (decrease) of at least 2-points in the weekly symptom scores for nausea at each of the last 6 weeks of the 12-week Treatment Period. Nausea was one of the items of the DGSSD assessed daily and recorded in the e-diary by the participant using an 11-point ordinal scale where: 0=no nausea to 10=worst possible nausea.
Time Frame: Baseline (Day-14 to Day-1) to (Week 6 to Week 12)
Population: mITT Population included all randomized participants with ≥1 postbaseline assessment of DGSSD.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Relamorelin 10 μg
Number analyzed (Participants) | 164 | 165
percentage of participants | 34.1 | 29.7

4. Secondary Outcome: Percentage of Participants Meeting the Abdominal Pain Responder Criterion During Each of the Last 6 Weeks of the 12-week Treatment Period
Description: An Abdominal Pain Responder was defined as a participant with an improvement (decrease) of at least 2-points in the weekly symptom scores for abdominal pain at each of the last 6 weeks of the 12-week Treatment Period. Abdominal pain was one of the items of the DGSSD assessed daily and recorded in the e-diary by the participant using an 11-point ordinal scale where: 0=no abdominal pain to 10=the worst possible abdominal pain and was recorded in an e-diary.
Time Frame: Baseline (Day-14 to Day-1) to (Week 6 to Week 12)
Population: mITT Population included all randomized participants with ≥1 postbaseline assessment of DGSSD.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Relamorelin 10 μg
Number analyzed (Participants) | 164 | 165
percentage of participants | 28.0 | 27.9

5. Secondary Outcome: Percentage of Participants Meeting the Bloating Responder Criterion During Each of the Last 6 Weeks of the 12-week Treatment Period
Description: A Bloating Responder was defined as a participant with an improvement (decrease) of at least 2-points in the weekly symptom scores for bloating at each of the last 6 weeks of the 12-week Treatment Period. Bloating was one of the items of the DGSSD assessed daily and recorded by the participant in the e-diary using an 11-point ordinal scale where: 0=no bloating and 10=the worst possible bloating and was recorded in the e-diary.
Time Frame: Baseline (Day-14 to Day-1) to (Week 6 to Week 12)
Population: mITT Population included all randomized participants with ≥1 postbaseline assessment of DGSSD.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Relamorelin 10 μg
Number analyzed (Participants) | 164 | 165
percentage of participants | 26.2 | 27.9

6. Secondary Outcome: Percentage of Participants Meeting the Postprandial Fullness Responder Criterion During Each of the Last 6 Weeks of the 12-week Treatment Period
Description: A Postprandial Fullness Responder was defined as a participant with an improvement (decrease) of at least 2-points in the weekly symptom scores for Postprandial Fullness at each of the last 6 weeks of the 12-week Treatment Period. Postprandial Fullness was one of the items of the DGSSD assessed daily and recorded by the participant in the e-diary using an 11-point ordinal scale where: 0=no feeling of fullness until finishing a meal (best) to 10=feeling full after only a few bites (worst).
Time Frame: Baseline (Day-14 to Day-1) to (Week 6 to Week 12)
Population: mITT Population included all randomized participants with ≥1 postbaseline assessment of DGSSD.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Relamorelin 10 μg
Number analyzed (Participants) | 164 | 165
percentage of participants | 22.6 | 25.5

7. Secondary Outcome: Number of Participants Who Experienced One or More Treatment-Emergent Adverse Events (TEAE)
Description: An adverse event (AE) is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study treatment. A TEAE is an AE that begins or worsens after receiving study drug.
Time Frame: Up to approximately 16 weeks
Population: Safety Population included all participants who received ≥1 administration of double-blind study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Relamorelin 10 μg
Number analyzed (Participants) | 163 | 163
Participants | 68 | 70

8. Secondary Outcome: Number of Participants With Potential Clinically Significant (PCS) Clinical Laboratory Results
Description: Clinical Laboratory tests included Hematology, Chemistry and Urinalysis tests. The investigator determined if the results were clinically significant. Only those categories where at least 1 person had a non-PCS value at Baseline and met the PCS criterion at least once during postbaseline are reported.
Time Frame: Up to 12 weeks
Population: Safety Population included all participants who received ≥1 administration of double-blind study treatment. Number analyzed is the number of participants with non-PCS baseline values and at least one post-baseline assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Relamorelin 10 μg
Number analyzed (Participants) | 163 | 163
Participants
  Eosinophils Absolute Cell Count [10^9/liter(L)]: >3×Upper Limit of Normal Value (ULN): number analyzed (Participants) | 152 | 158
  Eosinophils Absolute Cell Count [10^9/liter(L)]: >3×Upper Limit of Normal Value (ULN) | 0 | 1
  Hematocrit (RATIO): <0.9×Lower Limit of Normal Value (LLN): number analyzed (Participants) | 145 | 157
  Hematocrit (RATIO): <0.9×Lower Limit of Normal Value (LLN) | 2 | 2
  Hemoglobin (g/L): <0.9×LLN: number analyzed (Participants) | 147 | 153
  Hemoglobin (g/L): <0.9×LLN | 10 | 4
  Lymphocytes Absolute Cell Count (10^9/L): >1.5×ULN: number analyzed (Participants) | 151 | 158
  Lymphocytes Absolute Cell Count (10^9/L): >1.5×ULN | 1 | 0
  Lymphocytes Absolute Cell Count (10^9/L): <0.8×LLN: number analyzed (Participants) | 151 | 158
  Lymphocytes Absolute Cell Count (10^9/L): <0.8×LLN | 2 | 1
  Mean Corpuscular Volume [femtoliter (fL)]: >1.1×ULN: number analyzed (Participants) | 151 | 158
  Mean Corpuscular Volume [femtoliter (fL)]: >1.1×ULN | 2 | 0
  Neutrophils Absolute Cell Count (10^9/L): >1.5×ULN: number analyzed (Participants) | 150 | 156
  Neutrophils Absolute Cell Count (10^9/L): >1.5×ULN | 0 | 1
  Neutrophils Absolute Cell Count (10^9/L): <0.8×LLN: number analyzed (Participants) | 150 | 156
  Neutrophils Absolute Cell Count (10^9/L): <0.8×LLN | 2 | 3
  Platelet Count (Thrombocytes) (10^9/L): >1.5×ULN: number analyzed (Participants) | 152 | 158
  Platelet Count (Thrombocytes) (10^9/L): >1.5×ULN | 0 | 1
  Red Blood Cell Count (10^12/L): >1.1×ULN: number analyzed (Participants) | 151 | 159
  Red Blood Cell Count (10^12/L): >1.1×ULN | 0 | 1
  Red Blood Cell Count (10^12/L): <0.9×LLN: number analyzed (Participants) | 151 | 159
  Red Blood Cell Count (10^12/L): <0.9×LLN | 1 | 1
  White Blood Cell Count (10^9/L): >1.5×ULN: number analyzed (Participants) | 152 | 159
  White Blood Cell Count (10^9/L): >1.5×ULN | 1 | 1
  Bicarbonate (HCO3) (mmol/L): >1.1×ULN: number analyzed (Participants) | 152 | 156
  Bicarbonate (HCO3) (mmol/L): >1.1×ULN | 3 | 1
  Bicarbonate (HCO3) (mmol/L): >0.9×LLN: number analyzed (Participants) | 152 | 156
  Bicarbonate (HCO3) (mmol/L): >0.9×LLN | 3 | 1
  Blood Urea Nitrogen [millimoles(mmol/L)]: >1.2×ULN: number analyzed (Participants) | 137 | 153
  Blood Urea Nitrogen [millimoles(mmol/L)]: >1.2×ULN | 11 | 11
  Calcium (mmol/L): <0.9×LLN: number analyzed (Participants) | 153 | 160
  Calcium (mmol/L): <0.9×LLN | 0 | 1
  Cholesterol, Total, Non-Fasting (mmol/L): number analyzed (Participants) | 151 | 158
  Cholesterol, Total, Non-Fasting (mmol/L) | 0 | 1
  Creatinine [micromoles(μmol/L)]: >1.3×ULN: number analyzed (Participants) | 141 | 149
  Creatinine [micromoles(μmol/L)]: >1.3×ULN | 7 | 8
  Glucose-Chemistry, Fasting (mmol/L): >2.5×ULN: number analyzed (Participants) | 141 | 148
  Glucose-Chemistry, Fasting (mmol/L): >2.5×ULN | 10 | 21
  Glucose-Chemistry, Fasting (mmol/L): <0.9×LLN: number analyzed (Participants) | 141 | 148
  Glucose-Chemistry, Fasting (mmol/L): <0.9×LLN | 3 | 1
  Glycohemoglobin A1C: Increase of >=0.5%: number analyzed (Participants) | 155 | 160
  Glycohemoglobin A1C: Increase of >=0.5% | 91 | 125
  Glycohemoglobin A1C: Increase of >=1%: number analyzed (Participants) | 155 | 160
  Glycohemoglobin A1C: Increase of >=1% | 91 | 124
  Phosphorus (mmol/L): >1.1×ULN: number analyzed (Participants) | 147 | 156
  Phosphorus (mmol/L): >1.1×ULN | 2 | 5
  Phosphorus (mmol/L): <0.9×LLN: number analyzed (Participants) | 147 | 156
  Phosphorus (mmol/L): <0.9×LLN | 0 | 1
  Triglycerides, Fasting (mmol/L): >=3×ULN: number analyzed (Participants) | 149 | 154
  Triglycerides, Fasting (mmol/L): >=3×ULN | 5 | 5
  Uric Acid (Urate) (μmol/L): >1.1×ULN: number analyzed (Participants) | 123 | 130
  Uric Acid (Urate) (μmol/L): >1.1×ULN | 10 | 18
  Uric Acid (Urate) (μmol/L): <0.9×LLN: number analyzed (Participants) | 123 | 130
  Uric Acid (Urate) (μmol/L): <0.9×LLN | 1 | 3

9. Secondary Outcome: Number of Participants With Clinically Meaningful Trends for Vital Signs
Description: Vital Signs included assessments of heart rate, respiratory rate, systolic and diastolic blood pressure, and body temperature. The investigator determined if the results were clinically significant.
Time Frame: Up to 12 weeks
Population: Safety Population included all participants who received ≥1 administration of double-blind study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Relamorelin 10 μg
Number analyzed (Participants) | 163 | 163
Participants | 0 | 0

10. Secondary Outcome: Number of Participants With Clinically Significant Abnormal Electrocardiogram (ECG) Results
Description: A standard 12-lead ECG was performed. The investigator determined if the abnormal results were clinically significant.
Time Frame: Up to 12 weeks
Population: Safety Population included all participants who received ≥1 administration of double-blind study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Relamorelin 10 μg
Number analyzed (Participants) | 163 | 163
Participants | 4 | 3

11. Secondary Outcome: Number of Participants With a ≥1% Increase in Glycosylated Hemoglobin A1c (HBA1c)
Description: HbA1c is also known as glycosylated hemoglobin. It is the concentration of glucose bound to hemoglobin as a percentage of the absolute maximum that can be bound.
Time Frame: Baseline (Day 1) up to 12 weeks
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Relamorelin 10 μg
Number analyzed (Participants) | 163 | 163
Participants
  Glycohemoglobin A1C: Increase of >=0.5%: number analyzed (Participants) | 155 | 160
  Glycohemoglobin A1C: Increase of >=0.5% | 91 | 125
  Glycohemoglobin A1C: Increase of >=1%: number analyzed (Participants) | 155 | 160
  Glycohemoglobin A1C: Increase of >=1% | 91 | 124

12. Secondary Outcome: Number of Participants With Anti-relamorelin Antibody Testing Results by Visit
Description: A blood sample was collected that was sent to a laboratory for an anti-relamorelin antibody screening test. A positive screening test was confirmed by an immunodepletion assay. The number of participants in each of the following categories are reported: Negative Screening Test, Positive Screening Test, Negative Confirmatory Test, and Positive Confirmatory Test at each time point.
Time Frame: Baseline (Day 1), Day 14, Day 28, Day 84, and End of Treatment (Up to Day 84)
Population: Safety Population included all participants who received ≥ 1 administration of double-blind study treatment (N=163 in the Relamorelin 10 μg arm). Anti-relamorelin antibody testing was only done for those participants who received treatment with relamorelin. Number analyzed is the number of participants with data available at the given timepoint. Due to a laboratory issue not all positive screening tests were confirmed.
Measure: Count of Participants; unit: Participants
Arm/Group | Relamorelin 10 μg
Number analyzed (Participants) | 163
Participants
  Screening Test (Baseline): number analyzed (Participants) | 149
  Screening Test (Baseline): Negative | 133
  Screening Test (Baseline): Positive | 16
  Confirmatory Test (Baseline): number analyzed (Participants) | 15
  Confirmatory Test (Baseline): Negative | 13
  Confirmatory Test (Baseline): Positive | 2
  Screening Test (Day 14): number analyzed (Participants) | 137
  Screening Test (Day 14): Negative | 124
  Screening Test (Day 14): Positive | 13
  Confirmatory Test (Day 14): number analyzed (Participants) | 13
  Confirmatory Test (Day 14): Negative | 13
  Confirmatory Test (Day 14): Positive | 0
  Screening Test (Day 28): number analyzed (Participants) | 131
  Screening Test (Day 28): Negative | 115
  Screening Test (Day 28): Positive | 16
  Confirmatory Test (Day 28): number analyzed (Participants) | 16
  Confirmatory Test (Day 28): Negative | 15
  Confirmatory Test (Day 28): Positive | 1
  Screening Test (Day 84): number analyzed (Participants) | 111
  Screening Test (Day 84): Negative | 95
  Screening Test (Day 84): Positive | 16
  Confirmatory Test (Day 84): number analyzed (Participants) | 15
  Confirmatory Test (Day 84): Negative | 14
  Confirmatory Test (Day 84): Positive | 1
  Screening Test (End of Treatment): number analyzed (Participants) | 15
  Screening Test (End of Treatment): Negative | 13
  Screening Test (End of Treatment): Positive | 2
  Confirmatory Test (End of Treatment): number analyzed (Participants) | 2
  Confirmatory Test (End of Treatment): Negative | 2
  Confirmatory Test (End of Treatment): Positive | 0
  Screening Test (Unscheduled): number analyzed (Participants) | 4
  Screening Test (Unscheduled): Negative | 2
  Screening Test (Unscheduled): Positive | 2
  Confirmatory Test (Unscheduled): number analyzed (Participants) | 2
  Confirmatory Test (Unscheduled): Negative | 1
  Confirmatory Test (Unscheduled): Positive | 1

ADVERSE EVENTS:
Time Frame: Up to approximately 16 weeks
Description: All-Cause Mortality is based on the Intent-to-treat (ITT) Population. Safety Population, all participants who received ≥1 administration of double-blind study treatment, was used to determine the number of participants at risk for Serious Adverse Events and Other Adverse Events.
Arm/Group | Placebo | Relamorelin 10 μg
All-Cause Mortality (participants affected / at risk) | 0/167 | 0/169
Serious Adverse Events (participants affected / at risk) | 15/163 | 16/163
Other Adverse Events (participants affected / at risk) | 9/163 | 9/163
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=163) | Relamorelin 10 μg (N=163)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 1
Angina unstable (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1
Colitis (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 1
Diabetic gastroparesis (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Pneumonia (Infections and infestations) | 3 | 2
Diverticulitis (Infections and infestations) | 0 | 2
Urinary tract infection (Infections and infestations) | 2 | 1
Acute sinusitis (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 2 | 0
Cystitis (Infections and infestations) | 1 | 0
Pyelonephritis acute (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 2
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0
Anticoagulation drug level above therapeutic (Investigations) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Vertebral wedging (Musculoskeletal and connective tissue disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 2 | 1
Diabetic nephropathy (Renal and urinary disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 1
Hypovolaemic shock (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=163) | Relamorelin 10 μg (N=163)
Hyperglycaemia (Metabolism and nutrition disorders) | 9 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2019-02-08): https://cdn.clinicaltrials.gov/large-docs/08/NCT03285308/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-17): https://cdn.clinicaltrials.gov/large-docs/08/NCT03285308/SAP_001.pdf